CLINICAL TRIAL: NCT00606723
Title: Allogenic Stem Cell Transplantation for Children, Adolescents and Young Adults With Relapsed or Refractory AML; Multi Center Therapy Concept
Brief Title: Allogenic Stem Cell Transplantation for Children, Adolescents and Young Adults With Relapsed or Refractory AML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML SCT-BFM 2007; 2007-004517-34 (EudraCT Number)
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: relapsed or refractory AML; in children, adolescents and young adults
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Group I: Relapsed AML-patients with blast cell reduction to <20% before the second course of induction therapy. These patients will receive conventional SCT.
  Group II: Patients with non response to frontline treatment of AML, patients with blast cells <20% before the second course of induction therapy who do not achieve a second remission and relapsed AML-patients with blast cells >=20% before the second course of induction therapy. If these patients have a matched donor (MSD/MD) they will receive SCT with "FLAMSA".
  Group III: Patients who are eligible for Group II but have no matched donor. These patients will receive SCT from a haploidentical donor.
  Interventions: Biological: Hematopoietic stem cells from bone marrow or peripheral blood

INTERVENTIONS:
Biological: Hematopoietic stem cells from bone marrow or peripheral blood — > = 2 x 10*8 nucleated cells (WBC)/kg body weight of the recipient or rather > = 4 x 10*6 nucleated CD34+ cells / kg body weight are required for engraftment. Suspension of stem cells is administered via intravenous infusion.

SUMMARY:
1. To evaluate whether stem cell transplantation from a matched sibling donor is equivalent to a matched unrelated donor in in a second complete remission of acute myeloid leukemia (AML).
2. To evaluate whether stem cell transplantation (SCT) after chemotherapy (FLAMSA-schema) increases survival compared to a threshold derived from historical data
3. To evaluate whether SCT from haploidentical donors for children having no matched donor will result in better survival with acceptable toxicity.

DETAILED DESCRIPTION:
Target variables:

* Treatment response
* Event Free Survival
* Leukemia Free Survival
* Graft Versus Host Disease
* Regimen related toxicity

ELIGIBILITY:
Inclusion Criteria:

* Aged between 0-21 years
* Patients suffering from either refractory de novo AML or relapsed AML or patients with very high risk AML in CR1
* In sexually active patients two reliable contraception methods are used. This includes every combination of a hormonal contraceptive (such as injection, transdermal patch, implant, cervical ring) or of an intrauterine device(IUD) with a barrier method (e.g. diaphragm, cervical cap, or condom) or with a spermicide.
* Written informed consent of patient, parents or legal guardians

Exclusion Criteria:

* Severe renal impairment (GFR < 30% predicted for age)
* Pregnant or lactating females
* Current participation in another clinical trial
* Patients ≥ 12 years old for Group 1 ("BuCyMel") (patients younger that 12 years continue to be included)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 154 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
To evaluate whether stem cell transplantation (SCT) from a matched sibling donor (MSD) is equivalent to a matched unrelated donor (MUD) in second complete remission (CR2). | day 100
To evaluate whether "FLAMSA" increases leukemia free survival (LFS) and overall survival (OS) as compared to a historic control group | day 100
To evaluate whether SCT from haploidentical donors for children having no matched donor will result in an acceptable toxicity profile and a better LFS as compared to historic controls. | day 100

SECONDARY OUTCOMES:
Prospective evaluation of event free survival (EFS), LFS, and OS after SCT from either a MSD or a MUD | day 100
To evaluate whether it is feasible to standardize transplantation procedures in children with AML within the AML-Berlin/Frankfurt/Münster (BFM) study network | day 100
Decrease of transplantation associated mortality by standardized donor selection criteria | day 100
To further evaluate the contribution of immunomediated effects for the treatment of children suffering from very high risk AML | day 100
Prospective evaluation of late toxicities | day 100 and year 5

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sauer, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (24):
- Austria (3):
  - Graz University Hospital, Graz
  - Innsbruck University Hospital, Innsbruck
  - St. Anna Children Hospital, Vienna
- Teaching Hospital Motol, Prague, Czechia
- Germany (20):
  - University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg University Hospital, Heidelberg, Baden-Wurttemberg
  - University Children's Hospital Tübingen, Tübingen, Baden-Wurttemberg
  - University Children's Hospital Ulm, Ulm, Baden-Wurttemberg
  - University Children's Hospital Erlangen-Nürnberg, Erlangen, Bavaria
  - Dr. von Haunersches Kinderspital, München, Bavaria
  - University Hospital Würzburg, Würzburg, Bavaria
  - J.W. Goethe University Hospital and Faculty of Medicine, Frankfurt am Main, Hesse
  - Gießen University Hospital, Giessen, Hesse
  - Hannover Medical School, Department of Paediatrics, Paediatric Hematology and Oncology, Hanover, Lower Saxony
  - University Hospital Greifswald, Greifswald, Mecklenburg-West Pomerania
  - Düsseldorf University Hospital, Düsseldorf, North Rhine-Westphalia
  - University Hospital Essen, Essen, North Rhine-Westphalia
  - Münster University Hospital, Münster, North Rhine-Westphalia
  - Carl Gustav Carus University Children's Hospital Dresden, Dresden, Saxony
  - University Children's Hospital Halle, Halle, Saxony-Anhalt
  - University Hospital Kiel, Kiel, Schleswig-Holstein
  - University Children's Hospital Jena, Jena, Thuringia
  - Charité Campus Rudolf Virchow Hospital, Berlin
  - Hamburg-Eppendorf University Hospital, Hamburg